CLINICAL TRIAL: NCT02661685
Title: An Immunotherapy for Metastatic Cancer Patients by Adoptive Transfer of Autologous IKDC-like Cells - Phase 1 Clinical Trial
Brief Title: Safety Study of Adoptive Transfer of Autologous IKDC-like Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Academia Sinica, Taiwan (Other)
Responsible Party: Principal Investigator, Ming-Shen Dai, Attending physician, National Defense Medical Center, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IKDC-001
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Neoplasm Metastasis
Keywords: Cancer immunotherapy; IFN-γ-producing killer dendritic cell-like cells; Natural killer cells
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: 3+3 statistics model
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous IKDC-like cell (Experimental): Received autologous IKDC-like cells
  Interventions: Biological: autologous IKDC-like cells

INTERVENTIONS:
Biological: autologous IKDC-like cells — Subject received autologous IKDC-like cells every 14 days

SUMMARY:
The purpose of this study is to determine the safety of adoptive transferring autologous IKDC-like cells

DETAILED DESCRIPTION:
Cancer immunosurveillance in mice and human protects the host from outgrowth of tumor cells. This may establish a sufficient rationale for cancer immunotherapy that aims to control or eradicate tumor by an induction of effective anti-tumor immunity. The interest in developing cancer immunotherapy has intensified by the recent trials results showing durable responses in approximately 20% of patients who received various kinds of immunotherapy including adoptive transfer of tumor-specific T cells, cancer vaccines, and T cell response checkpoint blockade inhibition. Discoveries to date, natural killer (NK) cell function positively associates with reduction of cancer risk and with better survival of gastrointestinal stromal tumor patients. Interferon-producing killer dendritic cells (IKDCs) are a subpopulation of NK cells discovered in the mouse spleen, which can lyse tumor cells and acquire antigen presentation cell (APC) activity. We found putative IKDCs in human peripheral blood mononuclear cells (PBMCs); meanwhile, we also developed a method to expand IKDC-like cells from murine bone marrow and human PBMC ex vivo. The expanded human IKDC-like cells are cytotoxic toward several human leukemia cell lines and are capable to activate allogeneic T cells. For the in vivo anti-tumor activity, we found that two transfers of syngeneic murine IKDC-like cells reduced tumor burden in B16/OVA and B16/F10 melanoma and Lewis lung carcinoma models, and enhanced interferon (IFN)-γ production by the splenocytes of the tumor-bearing mice. Moreover, six transfers of IKDC-like cell significantly prolonged the survival of mice bearing B16/F10 melanoma. Based on these preclinical results, we hypothesize anti-tumor activity of human IKDC-like cells. We thus propose a phase 1 clinical trial to assess the safety of autologous IKDC-like cell therapy in metastatic cancer patients for determination of the maximum tolerated dose, and to monitor the immune parameters in patients before and after the IKDC-like cell transfer to investigate the therapeutic mechanism and biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic/recurrent non-hematological cancer, stage IV at study entry.
* Age: 21-75 years.
* ECOG performance status 0-1.
* Patients must have at least one measurable lesion.
* Patients' disease must have failed at least one-line of standard chemotherapy/targeted therapy or other treatment in the metastatic setting.
* Patients' estimated life expectancy is more than 3 months.
* Patients who refuse chemotherapy, or who are physiologically unsuitable for chemotherapy or any other standard therapy per investigator's discretion will be considered eligible for this trial.
* Patients must have adequate bone marrow function, defined as WBC ≥ 3500/mm3, neutrophil ≥ 1500/mm3, lymphocyte ≥ 1,000/mm3, and platelet ≥ 100,000/mm3.
* Patients must have adequate liver and renal function, defined as serum alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 5 times normal, bilirubin ≤ 1.5 times normal range, and creatinine ≤ 1.5 times upper normal limit.
* All patients should have documentation of negative result of penicillin test.
* Women or men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent.

Exclusion Criteria:

* Subjects with metastatic cancer in disease progression (expected survival time < 3 months).
* Subjects who have had chemotherapy less than 4 weeks before the start of trial.
* Subjects who received IFN-γ or GM-CSF less than 4 weeks before the start of trial.
* Subjects who are HIV, HBV, or HCV positive.
* Patients who have central nervous system metastasis except for those whose CNS disease have been treated with radiotherapy (Disease-free > 6 months) and/or surgery and have been stable for at least two weeks.
* Patients who have active acute or chronic infection (at the discretion of the investigator).
* Pregnant or breast-nursing women.
* Patients who have active cardiac disease requiring therapy for failure, angina, arrhythmia, or infarction within the preceding 6 months (exception: any patient whose cardiac failure is compensated on medications).
* Subjects who have received corticosteroids or other immunosuppressive agents less than 4 weeks before starting trial.
* Subjects who have asthma and/or are on treatment for asthma.
* Subjects with history of autoimmune disease, such as lupus, multiple sclerosis, Ankylosing Spondylitis, Systemic Sclerosis.
* Subjects with a history of other systemic disease..
* History of neoplastic disease within the last 5 years except for carcinoma in situ of the cervix, superficial bladder cancer or basal/squamous cell carcinoma of the skin.
* Subjects who present with open wounds.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of subject with Grade 3 or above adverse events that received autologous IKDC-like cells, graded according to NCI-CTCAE v4.03 | Through study complete, an average about 1.5 years
  I. Safety is evaluated by assessment of does-limiting toxicity (DLT) according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.03 or above.
  II. DLT is defined as follows:
  * Any Grade 3 or above toxicity regarding general disorders or immune disorders defined by NCI-CTCAE is determined by the investigator to be possibly related in causality to the treatment.
  * Fever, chillness, flu-like symptoms, or infusion-related reactions of grade 3 or more are to be counted as DLT only if they remain at grade 3 or more for more than three days despite of adequate symptomatic medications..
  III. The maximum tolerated dose (MTD) of autologous IKDC-like cell will be determined via a 3+3 traditional design.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shen Dai, MD/PhD, Principal Investigator — Attending Physician
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smyth MJ, Thia KY, Street SE, Cretney E, Trapani JA, Taniguchi M, Kawano T, Pelikan SB, Crowe NY, Godfrey DI. Differential tumor surveillance by natural killer (NK) and NKT cells. J Exp Med. 2000 Feb 21;191(4):661-8. doi: 10.1084/jem.191.4.661. PMID 10684858
- [Background] Vesely MD, Kershaw MH, Schreiber RD, Smyth MJ. Natural innate and adaptive immunity to cancer. Annu Rev Immunol. 2011;29:235-71. doi: 10.1146/annurev-immunol-031210-101324. PMID 21219185
- [Background] Galon J, Angell HK, Bedognetti D, Marincola FM. The continuum of cancer immunosurveillance: prognostic, predictive, and mechanistic signatures. Immunity. 2013 Jul 25;39(1):11-26. doi: 10.1016/j.immuni.2013.07.008. PMID 23890060
- [Background] Fridman WH, Pages F, Sautes-Fridman C, Galon J. The immune contexture in human tumours: impact on clinical outcome. Nat Rev Cancer. 2012 Mar 15;12(4):298-306. doi: 10.1038/nrc3245. PMID 22419253
- [Background] Chen DS, Mellman I. Oncology meets immunology: the cancer-immunity cycle. Immunity. 2013 Jul 25;39(1):1-10. doi: 10.1016/j.immuni.2013.07.012. PMID 23890059
- [Background] Rosenberg SA, Yang JC, Sherry RM, Kammula US, Hughes MS, Phan GQ, Citrin DE, Restifo NP, Robbins PF, Wunderlich JR, Morton KE, Laurencot CM, Steinberg SM, White DE, Dudley ME. Durable complete responses in heavily pretreated patients with metastatic melanoma using T-cell transfer immunotherapy. Clin Cancer Res. 2011 Jul 1;17(13):4550-7. doi: 10.1158/1078-0432.CCR-11-0116. Epub 2011 Apr 15. PMID 21498393
- [Background] Kochenderfer JN, Rosenberg SA. Treating B-cell cancer with T cells expressing anti-CD19 chimeric antigen receptors. Nat Rev Clin Oncol. 2013 May;10(5):267-76. doi: 10.1038/nrclinonc.2013.46. Epub 2013 Apr 2. PMID 23546520
- [Background] Galluzzi L, Vacchelli E, Eggermont A, Fridman WH, Galon J, Sautes-Fridman C, Tartour E, Zitvogel L, Kroemer G. Trial Watch: Adoptive cell transfer immunotherapy. Oncoimmunology. 2012 May 1;1(3):306-315. doi: 10.4161/onci.19549. PMID 22737606
- [Background] Thanendrarajan S, Nowak M, Abken H, Schmidt-Wolf IG. Combining cytokine-induced killer cells with vaccination in cancer immunotherapy: more than one plus one? Leuk Res. 2011 Sep;35(9):1136-42. doi: 10.1016/j.leukres.2011.05.005. Epub 2011 Jun 8. PMID 21652069
- [Background] Rosenberg SA, Restifo NP, Yang JC, Morgan RA, Dudley ME. Adoptive cell transfer: a clinical path to effective cancer immunotherapy. Nat Rev Cancer. 2008 Apr;8(4):299-308. doi: 10.1038/nrc2355. PMID 18354418
- [Background] Imai K, Matsuyama S, Miyake S, Suga K, Nakachi K. Natural cytotoxic activity of peripheral-blood lymphocytes and cancer incidence: an 11-year follow-up study of a general population. Lancet. 2000 Nov 25;356(9244):1795-9. doi: 10.1016/S0140-6736(00)03231-1. PMID 11117911
- [Background] Menard C, Blay JY, Borg C, Michiels S, Ghiringhelli F, Robert C, Nonn C, Chaput N, Taieb J, Delahaye NF, Flament C, Emile JF, Le Cesne A, Zitvogel L. Natural killer cell IFN-gamma levels predict long-term survival with imatinib mesylate therapy in gastrointestinal stromal tumor-bearing patients. Cancer Res. 2009 Apr 15;69(8):3563-9. doi: 10.1158/0008-5472.CAN-08-3807. Epub 2009 Apr 7. PMID 19351841
- [Background] Rusakiewicz S, Semeraro M, Sarabi M, Desbois M, Locher C, Mendez R, Vimond N, Concha A, Garrido F, Isambert N, Chaigneau L, Le Brun-Ly V, Dubreuil P, Cremer I, Caignard A, Poirier-Colame V, Chaba K, Flament C, Halama N, Jager D, Eggermont A, Bonvalot S, Commo F, Terrier P, Opolon P, Emile JF, Coindre JM, Kroemer G, Chaput N, Le Cesne A, Blay JY, Zitvogel L. Immune infiltrates are prognostic factors in localized gastrointestinal stromal tumors. Cancer Res. 2013 Jun 15;73(12):3499-510. doi: 10.1158/0008-5472.CAN-13-0371. Epub 2013 Apr 16. PMID 23592754
- [Background] Duan X, Deng L, Chen X, Lu Y, Zhang Q, Zhang K, Hu Y, Zeng J, Sun W. Clinical significance of the immunostimulatory MHC class I chain-related molecule A and NKG2D receptor on NK cells in pancreatic cancer. Med Oncol. 2011 Jun;28(2):466-74. doi: 10.1007/s12032-010-9480-9. Epub 2010 Mar 31. PMID 20354827
- [Background] McGilvray RW, Eagle RA, Watson NF, Al-Attar A, Ball G, Jafferji I, Trowsdale J, Durrant LG. NKG2D ligand expression in human colorectal cancer reveals associations with prognosis and evidence for immunoediting. Clin Cancer Res. 2009 Nov 15;15(22):6993-7002. doi: 10.1158/1078-0432.CCR-09-0991. Epub 2009 Oct 27. PMID 19861434
- [Background] de Kruijf EM, Sajet A, van Nes JG, Putter H, Smit VT, Eagle RA, Jafferji I, Trowsdale J, Liefers GJ, van de Velde CJ, Kuppen PJ. NKG2D ligand tumor expression and association with clinical outcome in early breast cancer patients: an observational study. BMC Cancer. 2012 Jan 18;12:24. doi: 10.1186/1471-2407-12-24. PMID 22257486
- [Background] Mamessier E, Sylvain A, Thibult ML, Houvenaeghel G, Jacquemier J, Castellano R, Goncalves A, Andre P, Romagne F, Thibault G, Viens P, Birnbaum D, Bertucci F, Moretta A, Olive D. Human breast cancer cells enhance self tolerance by promoting evasion from NK cell antitumor immunity. J Clin Invest. 2011 Sep;121(9):3609-22. doi: 10.1172/JCI45816. Epub 2011 Aug 15. PMID 21841316
- [Background] Taieb J, Chaput N, Menard C, Apetoh L, Ullrich E, Bonmort M, Pequignot M, Casares N, Terme M, Flament C, Opolon P, Lecluse Y, Metivier D, Tomasello E, Vivier E, Ghiringhelli F, Martin F, Klatzmann D, Poynard T, Tursz T, Raposo G, Yagita H, Ryffel B, Kroemer G, Zitvogel L. A novel dendritic cell subset involved in tumor immunosurveillance. Nat Med. 2006 Feb;12(2):214-9. doi: 10.1038/nm1356. Epub 2006 Jan 29. PMID 16444265
- [Background] Chan CW, Crafton E, Fan HN, Flook J, Yoshimura K, Skarica M, Brockstedt D, Dubensky TW, Stins MF, Lanier LL, Pardoll DM, Housseau F. Interferon-producing killer dendritic cells provide a link between innate and adaptive immunity. Nat Med. 2006 Feb;12(2):207-13. doi: 10.1038/nm1352. Epub 2006 Jan 29. PMID 16444266
- [Background] Himoudi N, Yan M, Bouma G, Morgenstern D, Wallace R, Seddon B, Buddle J, Eddaoudi A, Howe SJ, Cooper N, Anderson J. Migratory and antigen presentation functions of IFN-producing killer dendritic cells. Cancer Res. 2009 Aug 15;69(16):6598-606. doi: 10.1158/0008-5472.CAN-09-0501. Epub 2009 Aug 4. PMID 19654308
- [Background] Pletneva M, Fan H, Park JJ, Radojcic V, Jie C, Yu Y, Chan C, Redwood A, Pardoll D, Housseau F. IFN-producing killer dendritic cells are antigen-presenting cells endowed with T-cell cross-priming capacity. Cancer Res. 2009 Aug 15;69(16):6607-14. doi: 10.1158/0008-5472.CAN-09-0508. PMID 19679552
- [Background] Terme M, Mignot G, Ullrich E, Bonmort M, Minard-Colin V, Jacquet A, Schultze JL, Kroemer G, Leclerc C, Chaput N, Zitvogel L. The dendritic cell-like functions of IFN-producing killer dendritic cells reside in the CD11b+ subset and are licensed by tumor cells. Cancer Res. 2009 Aug 15;69(16):6590-7. doi: 10.1158/0008-5472.CAN-08-4473. PMID 19679551
- [Background] Chaudhry UI, Plitas G, Burt BM, Kingham TP, Raab JR, DeMatteo RP. NK dendritic cells expanded in IL-15 exhibit antitumor responses in vivo. J Immunol. 2007 Oct 1;179(7):4654-60. doi: 10.4049/jimmunol.179.7.4654. PMID 17878363
- [Background] Himoudi N, Nabarro S, Buddle J, Eddaoudi A, Thrasher AJ, Anderson J. Bone marrow-derived IFN-producing killer dendritic cells account for the tumoricidal activity of unpulsed dendritic cells. J Immunol. 2008 Nov 1;181(9):6654-63. doi: 10.4049/jimmunol.181.9.6654. PMID 18941256
- [Background] Liao N, Lee G, Chang C: Generation of murine and human interferon-producing killer cell-like cells with anti-tumor activity. . (patent pending) 2013.
- [Background] Lanier LL, Phillips JH, Hackett J Jr, Tutt M, Kumar V. Natural killer cells: definition of a cell type rather than a function. J Immunol. 1986 Nov 1;137(9):2735-9. No abstract available. PMID 3489775
- [Background] Burt BM, Plitas G, Nguyen HM, Stableford JA, Bamboat ZM, Dematteo RP. Circulating HLA-DR(+) natural killer cells have potent lytic ability and weak antigen-presenting cell function. Hum Immunol. 2008 Aug;69(8):469-74. doi: 10.1016/j.humimm.2008.06.009. Epub 2008 Jul 18. PMID 18640163
- [Background] Reagan-Shaw S, Nihal M, Ahmad N. Dose translation from animal to human studies revisited. FASEB J. 2008 Mar;22(3):659-61. doi: 10.1096/fj.07-9574LSF. Epub 2007 Oct 17. PMID 17942826
- [Background] Krause SW, Gastpar R, Andreesen R, Gross C, Ullrich H, Thonigs G, Pfister K, Multhoff G. Treatment of colon and lung cancer patients with ex vivo heat shock protein 70-peptide-activated, autologous natural killer cells: a clinical phase i trial. Clin Cancer Res. 2004 Jun 1;10(11):3699-707. doi: 10.1158/1078-0432.CCR-03-0683. PMID 15173076
- [Background] Ishikawa E, Tsuboi K, Saijo K, Harada H, Takano S, Nose T, Ohno T. Autologous natural killer cell therapy for human recurrent malignant glioma. Anticancer Res. 2004 May-Jun;24(3b):1861-71. PMID 15274367
- [Background] Parkhurst MR, Riley JP, Dudley ME, Rosenberg SA. Adoptive transfer of autologous natural killer cells leads to high levels of circulating natural killer cells but does not mediate tumor regression. Clin Cancer Res. 2011 Oct 1;17(19):6287-97. doi: 10.1158/1078-0432.CCR-11-1347. Epub 2011 Aug 15. PMID 21844012
- [Background] Yang YJ, Park JC, Kim HK, Kang JH, Park SY. A trial of autologous ex vivo-expanded NK cell-enriched lymphocytes with docetaxel in patients with advanced non-small cell lung cancer as second- or third-line treatment: phase IIa study. Anticancer Res. 2013 May;33(5):2115-22. PMID 23645763
- [Background] Yamaguchi T, Bamba K, Kitayama A, Kuroiwa Y, Yoshimatsu K, Shimakawa T, Ogawa K, Sekine T, Shimizu N, Yamamoto K. Long-term intravenous administration of activated autologous lymphocytes for cancer patients does not induce antinuclear antibody and rheumatoid factor. Anticancer Res. 2004 Jul-Aug;24(4):2423-9. PMID 15330194
- [Background] Delyon J, Mateus C, Lefeuvre D, Lanoy E, Zitvogel L, Chaput N, Roy S, Eggermont AM, Routier E, Robert C. Experience in daily practice with ipilimumab for the treatment of patients with metastatic melanoma: an early increase in lymphocyte and eosinophil counts is associated with improved survival. Ann Oncol. 2013 Jun;24(6):1697-703. doi: 10.1093/annonc/mdt027. Epub 2013 Feb 24. PMID 23439861
- [Background] Ku GY, Yuan J, Page DB, Schroeder SE, Panageas KS, Carvajal RD, Chapman PB, Schwartz GK, Allison JP, Wolchok JD. Single-institution experience with ipilimumab in advanced melanoma patients in the compassionate use setting: lymphocyte count after 2 doses correlates with survival. Cancer. 2010 Apr 1;116(7):1767-75. doi: 10.1002/cncr.24951. PMID 20143434
- [Background] Carthon BC, Wolchok JD, Yuan J, Kamat A, Ng Tang DS, Sun J, Ku G, Troncoso P, Logothetis CJ, Allison JP, Sharma P. Preoperative CTLA-4 blockade: tolerability and immune monitoring in the setting of a presurgical clinical trial. Clin Cancer Res. 2010 May 15;16(10):2861-71. doi: 10.1158/1078-0432.CCR-10-0569. Epub 2010 May 11. PMID 20460488
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867